CLINICAL TRIAL: NCT06624956
Title: Prevention and Treatment of Common Hyperglycemia in Surgery (PATCHS): A Randomized, Controlled, Pilot Study
Brief Title: Prevention and Treatment of Common Hyperglycemia in Surgery
Acronym: PATCHS
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, David Flum, Professor, Division of General Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00019463
Record Dates: First submitted 2024-09-25; First posted 2024-10-03 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-09

CONDITIONS: Surgery; Non Diabetic Hyperglycemia
MeSH Terms: interventions — Glucose; Insulin; Potassium

STUDY DESIGN:
Intervention Model Description: Potentially eligible patients will be approached on the day of surgery in a private room. Following formal, in person screening and informed consent by study team member who can thoroughly explain the study and answer patient questions, patients will be randomized to the study drug or to standard of care treatment (i.e. crystalloid infusion). All subjects will receive the same size bag of fluid and will have an infusion running during surgery. The administration of crystalloid is standard for surgeries performed at UW. Subjects in the standard/placebo arm will receive only regular crystalloid. Subjects in the GIK arm will receive regular crystalloid with GIK added. The contents of the bag will be blinded. The two fluids look the same to maintain blinding.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (Placebo Comparator): Subjects in the standard care/placebo arm will receive only regular crystalloid.
  Interventions: Drug: Crystalloid Infusion
- GIK (Active Comparator): Subjects in the glucose, insulin, and potassium (GIK) arm will receive regular crystalloid with GIK added.
  Interventions: Drug: glucose, insulin, and potassium (GIK); Drug: Crystalloid Infusion

INTERVENTIONS:
Drug: glucose, insulin, and potassium (GIK) — GIK formulation: 100 g/L glucose, 33 U/L insulin, and 40 mmol/L KCl
  Reference PMID: 32151220. Formulation represents a 50% reduction in compounded solute combination from the reference study, which allows for administration via peripheral IV.
  Arms: GIK
Drug: Crystalloid Infusion — placebo

SUMMARY:
The PATCH pilot trial aims to establish feasibility and determine the sample size of a future, large-scale, multi-site RCT, as well as reinforce the long-standing known safety profile of glucose, insulin, and potassium (GIK) and explore the physiologic response. We hypothesize that the use of GIK in non-diabetic patients undergoing abdominal surgery, will reduce rates of morbidity & death compared to standard of care treatment. In brief, primary outcomes of interest include estimation of the standard deviation (to derive a sample size estimation) and the ability to recruit target population, assessment of patient compliance/burden, and assessment of provider compliance/burden (feasibility).

DETAILED DESCRIPTION:
Elevated glucose levels during surgery are common and dramatically increase the risk of morbidity and mortality. This has been identified in multiple statewide quality improvement collaboratives, with a monotonic relationship between increased glucose levels and higher risks of almost all adverse events. While perioperative glucose management tends to focus on those with diabetes, some degree of perioperative hyperglycemia occurs in as much as two thirds of non-diabetic patients.

A recently identified phenomenon is that, at the same levels of hyperglycemia, non-diabetic patients have a much greater risk of death and complications compared to patients with diabetes. Given that hyperglycemia is typically considered a problem for people with diabetes, this finding has been described as a hyperglycemia paradox. Unfortunately, treatment with insulin can only happen after hyperglycemia has been recognized, and since non-diabetic patients are often not monitored for hyperglycemia, hyperglycemia is likely to be under-recognized. Moreover, addressing hyperglycemia after the fact may not be as effective in reducing adverse events as preventing hyperglycemia.

There is a long history of using perioperative insulin in patients undergoing at least one type of surgery. For over 45 years cardiac anesthesiologists have been testing the benefits of insulin combined with glucose and potassium (GIK) in cardiac surgery. In more than 30 RCTs, including more than 2000 patients with and without diabetes, GIK prophylaxis has been shown to be safe, with < 1 in 200 participants experiencing hypoglycemia secondary to the inclusion of glucose in the formulation. Moreover, these studies have found large reductions in surgically induced inflammation and often significant improvements in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older
2. Patients undergoing abdominal surgery planned to last greater than 4 hours with inpatient admission
3. Patients at UWMC - Montlake

3. Makes their own medical decisions: patient is deemed to have decisional capacity by the medical team and does not have a surrogate such as a spouse, partner, or caretaker making the decision on their behalf. Examples include patients with severe dementia or other cognitive limitations

Exclusion Criteria:

1. Known diagnosis of diabetes or altered glucose homeostasis during preoperative evaluation (single fasting blood sugar≥126 mg/dL or HbA1C≥6.5 percent).
2. Known diagnosis of chronic kidney disease (moderate-to-severe, or worse)

   * BMP within 6 months of screening is required. Patients with stage 3b (moderate-to-severe) kidney disease or worse (i.e. eGFR ≤ 30) will be excluded. Patients with a potassium reading greater than 5.5 at any point within the 6-month period will also be excluded.
3. Patients receiving chronic systemic steroids.
4. Patients undergoing cardiac or solid organ transplant procedures.
5. Surgery planned to last less than 4 hours.
6. Outpatient surgery
7. Pregnant people
8. Current UW Medicine or UW Dentistry residents and fellows
9. Known hypersensitivity to potassium, glucose, insulin, or any of its excipients.
10. Enrollment in another therapeutic study
11. Any serious underlying medical or psychiatric condition, dementia, altered mental status or any issue that would impair the ability of the patient to receive or tolerate the planned treatment, to understand informed consent or that in the opinion of the investigator would contraindicate the patient's participation in the study or that would confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
30-day Clinical NSQIP-defined serious adverse events | 30 days
  Estimate the standard deviation in support of anticipated, large-scale RCT for the outcome 30-day Clinical NSQIP-defined serious adverse events
Patient compliance/burden | 1 day
  Number patient refusal events vs enrolled
Ability to recruit the target population | 1 day
  Number of patients screened per month vs number of patients enrolled per month
Provider compliance/burden | 1
  Number of times GIK stopped for 20 minutes
Safety | 1 day
  Number of AEs and SAEs, thought to be at least possibly related to treatment, as well as associated AE type

SECONDARY OUTCOMES:
Number of hyperglycemic and hypoglycemic events | 1 day
  hyper- (BG>180) and hypoglycemic (BG <70)
Length of stay in hospital | 30 days
  Defined in post-op days

OTHER OUTCOMES:
Postoperative inflammation | 1 day
  Collect C-reactiev protein lab values
Postoperative inflammation | 1 day
  Collect blood cell count (CBC) lab values

CONTACTS AND LOCATIONS:
Overall Officials: David Flum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao K, Zhang Y, Li J, Cui Q, Zhao R, Chen W, Liu J, Zhao B, Wan Y, Ma XL, Yu S, Yi D, Gao F. Modified Glucose-Insulin-Potassium Regimen Provides Cardioprotection With Improved Tissue Perfusion in Patients Undergoing Cardiopulmonary Bypass Surgery. J Am Heart Assoc. 2020 Mar 17;9(6):e012376. doi: 10.1161/JAHA.119.012376. Epub 2020 Mar 10. PMID 32151220
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476